CLINICAL TRIAL: NCT04472507
Title: Use of Virtual Reality (VR) in Pain and Anxiety Reduction in Inpatient Paediatric Venepuncture and Cannulation
Brief Title: Virtual Reality for Children's Blood Sampling
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: B00823
Record Dates: First submitted 2020-07-02; First posted 2020-07-15 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Pain; Fear; Child, Only
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Virtual Reality (VR) is technology that simulates an immersive 3 dimensional environment for the user and is often used for immersive gaming experiences. The investigators will use VR in children who undergo painful procedures such as blood sampling and cannulation to investigate if VR reduces pain. The study will be carried out in 32 children admitted to the Royal Manchester Children in the UK and will assess feasbility of use VR, child and parent reported pain and therefore generate pilot data. This data will be used to design larger randomised control studies.

DETAILED DESCRIPTION:
Objectives

1. Conduct initial acceptability/feasibility testing of VRH use with children undergoing venepuncture or cannulation in an acute, often unplanned inpatient setting in a children's hospital.
2. Assess level of child and parent reported pain during procedure as well as change in heart rate.
3. Generate pilot data to design software and develop methods, outcome measures and patient/family engagement for a large randomised control trial (RCT) in the same setting to establish efficacy of VRH in reduction of perceived pain.

Outcome

1. Perceived and reported pain/anxiety scores for children undergoing venepuncture or cannulation with VRH.
2. Change in heart rate before, during and after painful procedure
3. Clinicians' feedback on the use of VRH in inpatient painful procedures

STUDY DESIGN and METHODS of DATA COLLECTION AND DATA ANALYIS Practitioners will be encouraged to contact the research team each time they are to perform a procedure between 0830H and 1600H and, unless already with another child using VRH, the research team will come to speak to parents to consent to the study. If consent is obtained then the procedure will be performed using current standard care as well as use of a VRH. The Oculus Go is a cheap and quick to set up headset. Off the shelf software will be selected that will distract but not require the movement of both arms. Software such as The Blu, Ocean Rift and Pet lab will be selected, dependent upon the age of the patient.

VRH will be brought to the room planned for procedure and set up for the child as part of the preparation for venepuncture/cannulation. Prior to application of VRH children will be asked to score their current pain score using the Wong Baker Faces Score (WBFS)1. This will be transcribed by the researcher. VRH use will be commenced at least 3 minutes prior to commencement of painful procedure. The procedure will then be performed by the practitioner and VRH supervised by parent(s). The researcher will not participate in the procedure beyond initial setup of the VRH to ensure real world feasibility is being tested for. Once the procedure is completed, the child will be allowed to continue using the VRH while clinicians and parents involved in the procedure fill in the feedback forms.

Feedback forms for parents will focus on perceived pain score and short qualitative review regarding acceptability, whether they would consider repeat application at subsequent venepuncture procedures, if VRH was well tolerated and whether they felt it helped. Feedback from clinicians will focus on ease of use of VRH, if they felt it facilitated procedure or whether it was felt to prolong the procedure. Forms will be filled in by parents and clinicians themselves and then handed to the researcher.

Children will then have the VRH removed and be asked to score their current pain again using the WBFS. Children's WBFS will be compared pre and post procedure. Assessment of acceptability/feasibility for children will be based on 3 questions - 1. Do they like it, 2. Was VRH wear comfortable and 3. Did they feel unwell whilst wearing VRH. Questionnaire answers will also be used to design future trials and bespoke VR software.

Questionnaires will then be pseudonymised and transcribed on to a secure computer for analysis of data. Interpretation of data will be performed by the clinical research team. Any statistical analysis required will be performed using SPSS Statistics 25 on pseydonymised datasets. Paper questionnaires will be kept in a locked drawer, in a locked room, on a locked research unit where access is only via swipe card. Access to paper questionnaires and digital data will only be for the immediate clinical research team of Professor Banerjee and Dr Worth.

1 Wong-Baker FACES Foundation (2018). Wong-Baker FACES® Pain Rating Scale. Retrieved [11/10/19}] with permission from http://www.WongBakerFACES.org

STUDY SETTING The study will be performed on all paediatric inpatient wards at Royal Manchester Hospital. The research team will be based on the CCRF (Children's Clinical Research Facility) and will move to each ward as required to provide VRH for procedures. Participants will be accessed via identification by clinicians performing painful procedures.

Royal Manchester Children's Hospital is the busiest children's hospital in the UK. Venepuncture and cannulation are routinely performed by a wide variety of staff including doctors, nurses and the IV access team. It is therefore an ideal location to conduct this study. Participants will undergo recruitment, discussion with the research team, consent and procedure all in the same location within Royal Manchester Children's Hospital. Participation in the study will not impact upon patient care and will not require patients or parents to move anywhere or do anything they would not already be doing as part of their inpatient stay.

Inclusion criteria Any child of age 5-12 years who are an inpatient in Royal Manchester Children's Hospital over a 4 week study period will be considered for consent if they require venepuncture or cannulation for a medical reason as determined by their lead medical team.

All individuals will be considered for inclusion in this study regardless of age, disability, gender reassignment, marriage and civil partnership, pregnancy and maternity, race, religion and belief, sex, and sexual orientation except where the study inclusion and exclusion criteria EXPLICITLY state otherwise.

Exclusion criteria Children under the age of 5 years (may not fit the headset, may become upset) and over the age of 12 years (pubertal, more mature understanding and expectations) will be excluded.

Children not needed venepuncture or cannulation will not be invited.

Children who have worn VRH previously and recognise dizziness/sickness or other ill health symptoms will not be asked to consent.

Parent/ guardians of children who are unsure about VRH will be excluded.

Parents will not be excluded if their first language is not English. As far as possible a translator will be arranged to translate child/parent responses and give feedback.

Size of sample For this feasibility study, the investigators aim to recruit 32 children during a 4 week period. Using the primary outcome acceptability of patient use, 32 children will enable us to identify our acceptability target of 75% of patients with 95% CI 56.6-88.5% (Clopper-Pearson exact). This number will also provide meaningful representation of a spread of gender, age groups, complexity of underlying illness, cultural and ethnic backgrounds to design future studies.

Recruitment The study will be advertised a month and two weeks prior to the start via email targeting all doctors, IV practitioners and nurses within Royal Manchester Children's Hospital informing them of the availability of VRH headsets for distraction during venepuncture/cannulation. Posters detailing similar information will be distributed across all paediatric wards and in treatment rooms. Information will also be available on the trust intranet.

Consent Informed consent will be taken from parents of patients recruited to the study. Both patients and parents will be given a written information sheet to read prior to consent. Once they have read this they will have the opportunity to ask any questions of the research team. If they agree to take part then parents will be asked to sign a consent form. Children will be given the option to sign an assent form if they wish but this will not be compulsory.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted as an inpatient in Royal Manchester Children's Hospital
* Patient requiring venepuncture or intravenous cannulation
* no specific medical diagnosis required for inclusion
* Child age 5-12 years during the study period

Exclusion Criteria:

* Child under the age of 5 years
* Child over the age of 12 years
* Child not requiring venepuncture or cannulation
* Child with previous discomofort wearing VRH

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children age 5-12 years, both males and females, can have any or no underlying condition, admitted to the Royal Manchester Children's Hospital and undergoing venepuncture or cannulation for clinical need.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
Perceived and reported pain/anxiety scores | Immediately before procedure
  Measures perceived and reported pain/anxiety scores for children undergoing venepuncture or cannulation with Virtual Reality Headsets. Wong Baker FACES Pain Rating Scale 0-10 will be used, with 0 representing "no hurt" and 10 "hurts worst".
Perceived and reported pain/anxiety scores | immediately following procedure
  Measures perceived and reported pain/anxiety scores for children undergoing venepuncture or cannulation with Virtual Reality Headsets. Wong Baker FACES Pain Rating Scale 0-10 will be used, with 0 representing "no hurt" and 10 "hurts worst".

SECONDARY OUTCOMES:
child heart rate before procedure | immediately prior to procedure
  heart rate measurement
Child heart rate during procedure | at any point during procedure
  heart rate measurement
Child heart rate after procedure | immediately following procedure
  heart rate measurement

OTHER OUTCOMES:
clinician feedback | immediately following procedure
  qualitative feedback following procedure

CONTACTS AND LOCATIONS:
Overall Officials: Indraneel Banerjee, Principal Investigator — Consultant Paediatric Endocrinologist
Locations (2):
- United Kingdom (2):
  - Indraneel Banerjee, Manchester
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No
high level data but not individual patient to be shared

REFERENCES:
- [Result] Ali S, McGrath T, Drendel AL. An Evidence-Based Approach to Minimizing Acute Procedural Pain in the Emergency Department and Beyond. Pediatr Emerg Care. 2016 Jan;32(1):36-42; quiz 43-4. doi: 10.1097/PEC.0000000000000669. PMID 26720064
- [Result] Chan E, Hovenden M, Ramage E, Ling N, Pham JH, Rahim A, Lam C, Liu L, Foster S, Sambell R, Jeyachanthiran K, Crock C, Stock A, Hopper SM, Cohen S, Davidson A, Plummer K, Mills E, Craig SS, Deng G, Leong P. Virtual Reality for Pediatric Needle Procedural Pain: Two Randomized Clinical Trials. J Pediatr. 2019 Jun;209:160-167.e4. doi: 10.1016/j.jpeds.2019.02.034. Epub 2019 Apr 29. PMID 31047650

DOCUMENTS (1):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT04472507/Prot_000.pdf